CLINICAL TRIAL: NCT00925184
Title: Students' View: Survey of Medical Education in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Wing Pong Chan, Taipei Medical University-Wanfang Hospital
Other Study IDs: WF-R-CWP-97-001
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Understand Students' View Toward Current Medical Education.
Keywords: questionnaire, medical education, medical students.

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- medical students, graduate year,: medical students at graduate year will be invited to participate in this study.

SUMMARY:
The aim of this research project is to establish a students' perspective to most medical schools in Taiwan. We expect that these surveys will provide helpful information to candidates for selection of medical school before admission, and will also be a useful reference guide to improve quality of medical education to our governmental policy makers.

DETAILED DESCRIPTION:
The aim of this research project is to establish a students' perspective to most medical schools in Taiwan. We will select Medical School Graduation Questionnaires, obtained from Association of American Medical Colleges, AAMC, which has been performed in US for more than 30 years. These questionnaires will modify with edition with expert opinions of our country. We will invite students' representative of each school for survey visit and deliver questionnaires to students after complete communication and permission of their schools. These surveys include learning resources, student support services, student daily life, medical education…etc. We expect that these surveys will provide helpful information to candidates for selection of medical school before admission, and will also be a useful reference guide to improve quality of medical education to our governmental policy makers.

ELIGIBILITY:
Inclusion Criteria:

* medical students at their graduate year and are willing to fill out the questionnaire.

Exclusion Criteria:

* medical students who do not want to fill out the questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical students at their graduate year will be invited to participated in this study. students who are willing to participate need to help us to fill out a questionnaire about their educational experience in medical school.
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Filled out the assigned questionnaire. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Wing Pong Chan, MD, Principal Investigator — Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wanfang Hospital, Taipei, Taiwan